CLINICAL TRIAL: NCT06603623
Title: Phase 2 Double-Blind, Randomized, Placebo Controlled, Efficacy and Safety Trial of BHV-2100 for the Acute Treatment of Migraine
Brief Title: Efficacy and Safety Trial of BHV-2100 for the Acute Treatment of Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biohaven Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Organization: Biohaven Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV2100-201
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Migraine
Keywords: Acute Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BHV-2100 75 mg (Experimental)
  Interventions: Drug: BHV-2100
- BHV-2100 150 mg (Experimental)
  Interventions: Drug: BHV-2100
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BHV-2100 — BHV-2100 75mg
  Arms: BHV-2100 75 mg
Drug: BHV-2100 — BHV-2100 150 mg
  Arms: BHV-2100 150 mg
Drug: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
This study is designed to identify at least one dose of BHV-2100 that is safe and effective in reducing headache pain and other symptoms in the treatment of migraine.

ELIGIBILITY:
Key Inclusion Criteria:

Participants with at least 1 year history of migraine (with or without aura) consistent with a diagnosis according to the International Classification of Headache Disorders, 3rd Edition,19 including the following:

1. 2-8 migraine headache attacks of moderate or severe intensity in each of the 3 months prior to the Screening Visit and throughout the Screening Period.
2. Less than 15 days with headaches (migraine or non-migraine) per month in each of the 3 months prior to the Screening Visit and throughout the Screening Period.
3. Participants on prophylactic migraine medication are permitted to remain on therapy they have been on a stable dose for at least 3 months prior to the Screening Visit.

Key Exclusion Criteria:

1. Participants with a history of basilar migraine or hemiplegic migraine.
2. Participants who have taken medication for acute treatment of headache (including triptans, ergotamine, opioids, acetaminophen, NSAIDs, or combination analgesics) on 10 or more days in any of the 3 months prior to screening.
3. Participants who have used a neuromodulation device for migraine treatment over the preceding 3 months before screening.
4. History of chronic active infection (e.g., HIV, hepatitis B or C, tuberculosis, etc.), or individuals who have received anti-HCV treatment within 6 months prior to Screening.
5. Participant history with current evidence of uncontrolled, unstable or recently diagnosed cardiovascular disease, such as ischemic heart disease, coronary artery vasospasm, and cerebral ischemia. participants with Myocardial Infarction (MI), Acute Coronary Syndrome (ACS), Percutaneous Coronary Intervention (PCI), cardiac surgery, stroke or transient ischemic attack (TIA) during the 6 months prior to screening.
6. Uncontrolled hypertension (high blood pressure), or uncontrolled diabetes (however, participants can be included who have stable hypertension and/or stable diabetes for at least 3 months prior to being enrolled). A single blood pressure measurement of greater than 150 mm Hg systolic or 100 mm Hg diastolic after 10 minutes of rest is exclusionary.
7. Participant has a current diagnosis of major depression, other pain syndromes (e.g. chronic pelvic pain, chronic regional pain syndrome, fibromyalgia), psychiatric conditions (e.g., schizophrenia), dementia, or significant neurological disorders (other than migraine) that, in the Investigator's opinion, might interfere with study assessments.
8. Participant has a history of gastric, or small intestinal surgery (including gastric bypass, gastric banding, gastric sleeve, gastric balloon, etc.), or other disease or condition (e.g. chronic pancreatitis, ulcerative colitis, etc.) that causes malabsorption.
9. Participant is on or has a recent history (past 30 days) of concomitant use of moderate/strong CYP3A4 inhibitors or inducers.
10. Participant is on or has a recent history (past 30 days) of concomitant use of moderate/strong p-gp or BCRP inhibitors.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 647 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Freedom From Pain at 2 Hours Post-dose | 2 hours post-dose
  Pain levels are assessed on a 4-point scale (none, mild, moderate, severe) using the electronic diary (eDiary). Pain freedom is defined as pain level of none. Coprimary endpoints will be tested hierarachically by dose
Percentage of Participants With Freedom From Most Bothersome Symptom (MBS) at 2 Hours Post-dose | 2 hours post-dose
  MBS is reported as nausea, photophobia, or phonophobia at migraine onset using the eDiary. Symptom status (absent, present) is assessed post-dose using the eDiary separately for nausea, photophobia, and phonophobia. Freedom from MBS is defined as MBS reported at onset that was absent post-dose. Coprimary endpoints will be tested hierarachically by dose

SECONDARY OUTCOMES:
Percentage of Participants With Pain Relief at 2 Hours Post-dose | 2 hours post-dose
  Pain levels are assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Pain relief is defined as pain level of none or mild.
Percentage of Participants With Return to Normal Function at 2 Hours Post-dose | 2 hours post-dose
  Return to normal function at 2 hours post-dose is assessed using the percentage of subjects with a functional disability level of normal at 2 hours post-dose in the subset of subjects with functional disability at the time of dosing. Functional disability level is measured on a 4-point numeric rating scale (0=normal, 1=mildly impaired, 2=severely impaired, 3=requires bedrest), and functional disability is defined as mildly impaired, severely impaired, or requires bedrest.
Percentage of Participants With Sustained Pain Relief From 2 to 24 Hours Post-dose | From 2 hours up to 24 hours post-dose
  Pain levels are assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Sustained pain relief is defined as pain level of none or mild at 2 hours up to 24 hours post-dose with no rescue medication use through 24 hours post-dose.
Percentage of Participants With Sustained Pain Relief From 2 to 48 Hours Post-dose | From 2 hours up to 48 hours post-dose
  Pain levels are assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Sustained pain relief is defined as pain level of none or mild at 2 hours up to 48 hours post-dose with no rescue medication use through 48 hours post-dose.
Percentage of Participants With Sustained Pain Freedom From 2 to 24 Hours Post-dose | From 2 hours up to 24 hours post-dose
  Pain levels are assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Sustained pain freedom is defined as pain level of none at 2 hours up to 24 hours post-dose with no rescue medication use through 24 hours post-dose.
Percentage of Participants With Sustained Pain Freedom From 2 to 48 Hours Post-dose | From 2 hours up to 48 hours post-dose
  Pain levels are assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Sustained pain freedom is defined as pain level of none at 2 hours up to 48 hours post-dose with no rescue medication use through 48 hours post-dose.
Percentage of Participants With Freedom From Phonophobia at 2 Hours Post-dose | 2 hours post-dose
  Phonophobia (sensitivity to sound) status is measured as absent 2 hours postdose in the subset of subjects with phonophobia present at the time of dosing in the eDiary. Freedom from phonophobia is defined as phonophobia absent.
Percentage of Participants With Freedom From Photophobia at 2 Hours Post-dose | 2 hours post-dose
  Photophobia (sensitivity to light) status is measured as absent 2 hours postdose in the subset of subjects with photophobia present at the time of dosing in the eDiary. Freedom from photophobia is defined as photophobia absent.
Percentage of Participants With Rescue Medication Use Within 24 Hours Post-dose | 24 hours post-dose
  Participants who do not experience relief of their migraine headache at the end of 2 hours after dosing with study medication (and after the 2-hour assessments has been completed on the eDiary) are permitted to use the following rescue medications: aspirin, ibuprofen, acetaminophen up to 1000 mg/day (this includes Excedrin Migraine), naproxen (or any other type of nonsteroidal anti-inflammatory drug), antiemetics (e.g., metoclopramide or promethazine), or baclofen. The participant's use of rescue medication is recorded by the participant in a paper diary.
Percentage of Participants With Freedom From Nausea at 2 Hours Post-dose | 2 hours post-dose
  Nausea status is measured as absent 2 hours postdose in the subset of subjects with nausea present at the time of dosing in the eDiary. Freedom from nausea is defined as nausea absent.
Percentage of Participants With Pain Relapse From 2 to 48 Hours Post-dose | From 2 hours up to 48 hours post-dose
  Pain levels are assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Pain relapse is defined as pain level of mild, moderate, or severe after 2 hours up to 48 hours for the participants who are pain-free at 2 hours post-dose.
Observed Plasma concentration in Patients After a Single Dose of BHV-2100 | At 2, 8, and 24 hours post-dose
Number of Participants with Deaths, Serious AEs (SAEs), and moderate or severe AEs | Up to 11 weeks
  To assess the tolerability and safety of BHV-2100. This objective will be measured by assessing the number of unique subjects with deaths, SAEs, and moderate and severe AEs.
Number of Subjects with Clinically Significant Laboratory Abnormalities | Up to 11 weeks
  To assess the tolerability and safety of BHV-2100. This objective will be measured by assessing the number of unique subjects with grade 3 and 4 laboratory abnormalities.

CONTACTS AND LOCATIONS:
Locations (60):
- United States (60):
  - MD First Research, Gilbert, Arizona
  - WR-PRI, LLC (Encino), Encino, California
  - Cenexel CNS Los Alamitos, Los Alamitos, California
  - Clinical Research Institute, Los Angeles, California
  - WR-PRI, LLC (Newport Beach), Newport Beach, California
  - Cenexel CIT IE, Riverside, California
  - Hasbani Neurology, New Haven, Connecticut
  - Ki Health Partners DBA/ New England Institute for Clinical Research, Stamford, Connecticut
  - Green Leaf Clinical Trials, Jacksonville, Florida
  - WR-MSRA (Multi-Specialty Research Associates), Lake City, Florida
  - AppleMed Research Group, Miami, Florida
  - Ideal Research, Pembroke Pines, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Premier Research Instiute, West Palm Beach, Florida
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Velocity Clinical Research, Savannah, Savannah, Georgia
  - Chicago Headache Center & Research Center, Chicago, Illinois
  - Healthcare Research Network II, LLC, Flossmoor, Illinois
  - Velocity Clinical Research, Sioux City, Sioux City, Iowa
  - Integrated Clinical Trials Services, West Des Moines, Iowa
  - Collective Medical Research, Overland Park, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Crescent City Headache & Neurology, Chalmette, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Velocity Clinical Research, Rockville, Rockville, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Neurology Center of New England PC, Foxborough, Massachusetts
  - MedVadis Research Corp, Waltham, Massachusetts
  - Mass Institute of Clinical Research, Westborough, Massachusetts
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Quest Research Institute, Farmington Hills, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - StudyMedrix Research, City of Saint Peters, Missouri
  - Alliance for Multispecialty Research - Kansas City, Kansas City, Missouri
  - Clinvest Research, Springfield, Missouri
  - WR-CRNC (Wake Research), Las Vegas, Nevada
  - ActivMed Practices & Research-Portsmouth/Pease, Portsmouth, New Hampshire
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Fieve Clinical Research, Inc., New York, New York
  - Rochester Clinical Research, Rochester, New York
  - Velocity Clinical Research, Vestal, Vestal, New York
  - PharmQuest Life Sciences, Greensboro, North Carolina
  - Accellacare of Raleigh, Raleigh, North Carolina
  - Hometown Urgent Care and Research, Dayton, Ohio
  - OK Clinical Research, LLC, Edmond, Oklahoma
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Velocity Clinical Research, Columbia, Columbia, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - KCA Neurology, Franklin, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - Zenos Clinical Research, Dallas, Texas
  - DM Clinical Research - Belliare, Houston, Texas
  - Red Star Research, LLC, Lake Jackson, Texas
  - Epic Clinical Research, Lewisville, Texas
  - DM Clinical Research - Tomball, Tomball, Texas
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Seattle Clinical Research Center, Seattle, Washington